CLINICAL TRIAL: NCT01215981
Title: MT2010-08R Influenza Vaccine Specific Immune Responses After Allogeneic Hematopoietic Cell Transplantation: Are One or Two Vaccine Doses Needed?
Brief Title: Influenza Vaccine Post Allogeneic Transplant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patients and no longer influenza vaccine season.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010NTLS050; MT2010-08R (Other: Blood and Bone Marrow Transplantation Program); 1007M86296 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Results first posted 2016-08-16 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Hematopoietic Stem Cell Transplant; Hematologic Malignancy
Keywords: influenza vaccine
MeSH Terms: conditions — Hematologic Neoplasms; Influenza, Human | interventions — Influenza Vaccines; Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Participants Receiving 1 Dose of Vaccine (Active Comparator): Control group participants (healthy volunteers):
  * Age 18 to 50 years
  * No history of previous allergic reaction to influenza vaccine, known egg allergy or Guillan-Barre Syndrome
  * No flu vaccine in previous 4 months
  and/or HSCT recipients who are greater than 60 days post transplant.
  Interventions: Biological: Influenza vaccine
- Participants Receiving 2 Doses of Vaccine (Active Comparator): Hematopoietic stem cell transplant (HSCT) recipients who are greater than 60 days post transplant.
  Interventions: Biological: Influenza vaccine

INTERVENTIONS:
Biological: Influenza vaccine — One dose of inactivated hemagglutinins of influenza A (H1N1, H3N2) and influenza B
  Other Names: H1N1; H3N2; Influenza A vaccine; Influenza B vaccine
  Arms: Participants Receiving 1 Dose of Vaccine
Biological: Influenza vaccine — Two doses of inactivated hemagglutinins of influenza A (H1N1, H3N2) and influenza B
  Other Names: Influenza A; H1N1; N3N2; Influenza B
  Arms: Participants Receiving 2 Doses of Vaccine

SUMMARY:
Study Design:

This is a randomized, single center study to evaluate immune responses to the seasonal influenza vaccine in allogeneic hematopoietic stem cell transplant (HSCT) recipients who receive one vaccine or two vaccine doses one month apart. In addition, a cohort of healthy adult volunteers will be recruited as controls to confirm immune response to a single influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Patient Population

  * HSCT recipients who are greater than 60 days post transplant.
  * Age 6 months and older who are greater than 60 days post post allogeneic hematopoietic cell transplant
  * Show neutrophil recovery, platelet count > 50,000/mm3 (may be transfused), no known disease relapse
  * No history of previous allergic reaction to influenza vaccine, known egg allergy or Guillan-Barre Syndrome
  * No flu vaccine in previous 4 months, no Campath in previous 6 months, no intravenous immune globulin (IVIG) in previous 3 months
* Controls:

  * Age 18 to 50 years
  * No history of previous allergic reaction to influenza vaccine, known egg allergy or Guillan-Barre Syndrome
  * No flu vaccine in previous 4 months

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Verneris, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- See also: Randomized Trial of One versus Two Doses of Influenza Vaccine after Allogeneic Transplantation — http://dx.doi.org/10.1016/j.bbmt.2012.08.015

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The original study design included healthy adult volunteers in addition to the HSCT recipients; however, the protocol was modified to exclude the healthy volunteers.
Period: Overall Study
Arm/Group | HSCT Recipients Who Were Randomized to 1 Vaccine Dose | HSCT Recipients Who Were Randomized to 2 Vaccine Doses
Started | 35 | 33
Completed | 33 | 32
Not Completed | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HSCT Recipients Who Were Randomized to 1 Vaccine Dose | HSCT Recipients Who Were Randomized to 2 Vaccine Doses | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 9 | 17
  Between 18 and 65 years | 25 | 22 | 47
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 19 | 19 | 38
Region of Enrollment [Number; unit: participants]
  United States | 33 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With T-Cell Based Immune Response to Vaccine
Description: The primary endpoint of this study is to measure the response to the vaccine with laboratory studies including viral specific T cell immune responses. Response is defined as 4 times above the background after a filter plate was developed. Response is listed as a number of subjects (evaluable) that successfully responded.
Time Frame: 8 Weeks After Vaccination
Population: One of the 33 participants randomized to receive 1 vaccine dose died prior to the 8 week evaluation.
Measure: Number; unit: Patients
Groups:
- HSCT Recipients Who Were Randomized to 1 Vaccine Dose: Allogeneic hematopoietic stem cell transplant (HSCT) recipients who received 1 dose (day of enrollment) of seasonal influenza vaccine after transplant.
- HSCT Recipients Who Were Randomized to 2 Vaccine Doses: Allogeneic hematopoietic stem cell transplant (HSCT) recipients who received 2 doses (day of enrollment and 4 weeks after later) of seasonal influenza vaccine after transplant.
Arm/Group | HSCT Recipients Who Were Randomized to 1 Vaccine Dose | HSCT Recipients Who Were Randomized to 2 Vaccine Doses
Number analyzed (Participants) | 32 | 32
Patients | 14 | 15

2. Secondary Outcome: Number of Subjects With H3 Based Immune Response to Vaccine
Description: The secondary endpoint of this study is to measure the response to the vaccine with laboratory studies including viral specific H3 immune responses (IFN-y Elispot). Response is defined as 4 fold increase in H3N1. Response is listed as a number of subjects (evaluable) that successfully responded.
Time Frame: 8 Weeks After Vaccination
Population: One of the 33 participants randomized to receive 1 vaccine dose died prior to the 8 week evaluation.
Measure: Number; unit: Patients
Arm/Group | HSCT Recipients Who Were Randomized to 1 Vaccine Dose | HSCT Recipients Who Were Randomized to 2 Vaccine Doses
Number analyzed (Participants) | 32 | 32
Patients | 4 | 7

ADVERSE EVENTS:
Arm/Group | HSCT Recipients Who Were Randomized to 1 Vaccine Dose | HSCT Recipients Who Were Randomized to 2 Vaccine Doses
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/33 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes